CLINICAL TRIAL: NCT02884570
Title: Post-hospital Evaluation of Anxiety / Depression in Parents of Children Who Required Tracheostomy Before the Age of 1 Year
Brief Title: Parental Mental Health After Tracheostomy in Early Childhood
Acronym: TRACH
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9253
Record Dates: First submitted 2016-08-04; First posted 2016-08-31 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Tracheotomised Children; Anxiety of Parents; Depression of Parents
Keywords: Tracheotomy; Anxiety; Depression; Back Home
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Auto-Questionnaires — Consents and questionnaires will be sent to the parental home or filled in an interview with an investigator (or telephone consultation).

SUMMARY:
To assess the prevalence of anxiety / depression in post- hospital for parents (mothers and fathers) of children with tracheotomy before the age of 1 year between 2000 and 2012.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the level of anxiety / depression of families and to correlate to the lived parental of tracheotomy and indirectly that of the child (hetero - evaluation).

The information from this study should allow staff to refine and adjust their practices in terms of information and support for families with tracheotomised children. The information given to families before the establishment of a tracheotomy for their child may also be adapted.

ELIGIBILITY:
Inclusion criteria :

Families whose child :

* Has been tracheotomised before the age of 1 year between 2000 and 2012
* Came out of hospital with a tracheotomy tube
* Is or has been followed by one of three centers

Exclusion criteria :

* Children decannulated before hospital discharge .
* Death before the start of the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents (mothers and fathers) of children with tracheotomy before the age of 1 year between 2000 and 2012.
  Pre- selection will take place in Pediatric Neonatal and Reanimation services of Montpellier, Paris (Hôpital Robert Debré ) and Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Anxiety and Depression | Through study completion, up to 6 months
  Auto-questionnaire Hospital Anxiety and Depression Scale HADS

SECONDARY OUTCOMES:
Experienced of the care by the families | Through study completion, up to 6 months
  Auto-questionnaire Hartnick

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Cambonie, Professor, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided